CLINICAL TRIAL: NCT02897908
Title: Non-invasive Liver Screening Using FibroScan Device for Liver Disease Patients for the Steatosis/Fibrosis Database
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Ajay Chaudhuri, Principal Investigator, State University of New York at Buffalo
Other Study IDs: FibroScan
Record Dates: First submitted 2016-09-03; First posted 2016-09-13 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Disease of Liver and Bile Duct
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver fibrosis and steatosis: measurements of liver fibrosis and steatosis will be obtained using Vibration controlled transient elastography FDA approved device- FibroScan for the purpose of building a data base of potential subjects for future research.
  Interventions: Procedure: vibration controlled transient elastography (VCTE)

INTERVENTIONS:
Procedure: vibration controlled transient elastography (VCTE) — Once on the examination table, the subject will be instructed to place the right arm under their head and to cross their right ankle over the left ankle. The subject will then be asked to slightly bend to the left side to open the intercostal space. Subsequently, a handheld probe is placed in the intercostal space overlaying the right hepatic lobe. The velocity of returning shear waves, measured at a depth of 25-65 mm, is converted into a liver stiffness measurement (LSM). The LSM obtained from a given VCTE exam is the median value of at least 10 successful measurements. This information, along with clinical data associated with the patient will be placed in a database for use in identifying potential subjects for future trials.
  Other Names: fibroscan

SUMMARY:
The primary goal of this study is to establish a database of people with varying levels of hepatic fibrosis and various etiologies of liver disease for use in future research protocols.

DETAILED DESCRIPTION:
The Fibroscan device will determine liver stiffness as well as the amount of fat through another application on the machine called controlled attenuation parameter or Controlled Attenuation Parameters (CAP). The liver stiffness measurements are then translated into a score that tells how much liver fibrosis or fat is present. Patients identified with potential for fatty liver or specific liver-related diseases causing fibrosis would be approached for a voluntary FibroScan measurement. From these patients, the investigators will collect information related to demographics, disease history, medical comorbidities, social history, laboratory and radiologic parameters. This information, along with clinical data associated with the patient will be placed in a database for use in identifying potential subjects for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known, or suspected risk factors for steatosis (fat) or hepatic fibrosis
* Subjects who have been previously diagnosed with Non-Alcoholic Steatohepatitis (NASH) but who do not have current steatosis (fat) or fibrosis scoring
* Subjects who have other known liver diseases ie: HCV

Exclusion Criteria:

* Patients less than 18 years of age
* Pregnancy
* Patients that do not want to be contacted for consideration in future research studies.
* Patients diagnosed with ascites or peritoneal dialysis
* Body mass index (BMI) ≥40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subjects with known, or suspected risk factors for steatosis (fat) or hepatic fibrosis
  * Subjects who have been previously diagnosed with Non-Alcoholic Steatohepatitis (NASH) but who do not have current steatosis (fat) or fibrosis scoring
  * Subjects who have other known liver diseases ie: hepatitis C virus (HCV)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
measurement of fibrosis in patients with varying degrees of liver disease | 10 years
  single event per patient with liver disease to measure degree of fibrosis concentration

SECONDARY OUTCOMES:
measurement of liver fat in patients with varying degrees of liver disease | 10 years
  single event per patient with liver disease to measure degree of fat concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Conventus Medical Office Building, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided